CLINICAL TRIAL: NCT02670408
Title: Diagnostic and Therapeutic Applications of Microarrays in Heart Transplantation, a Multicenter Study (INTERHEART)
Brief Title: Diagnostic and Therapeutic Applications of Microarrays in Heart Transplantation
Status: Recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Philip Halloran, Distinguished Professor, University of Alberta
Other Study IDs: ATAGC 002
Record Dates: First submitted 2016-01-22; First posted 2016-02-01 (Estimated); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Cardiac Transplant Disorder
Keywords: Heart transplant; global gene expression; molecular diagnostics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biopsy extract containing RNA
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Endomyocardial biopsy — One of several endomyocardial biopsy bites taken as the standard of care. We are asking now for two endomyocardial biopsy bites, to determine tissue sampling variability.

SUMMARY:
Demonstrate the impact of the Molecular Microscope Diagnostic System as the standard of care for heart transplant patients.

DETAILED DESCRIPTION:
The current standard for biopsy-based diagnoses of rejection of heart transplants is the ISHLT classification from 2004, which represents a widely-used international consensus, based on morphological criteria of the cellular infiltrate within the myocardial specimen system with certainties and some arbitrary and blurred parameters. Recent data-driven approaches using molecular and conventional technologies indicate that this system produces incorrect diagnoses with potential harm to patients due to inappropriate treatment. To address this unmet need and improve diagnostics in the area of organ transplantation, the Alberta Transplant Applied Genomics Centre (ATAGC, University of Alberta) has developed a new diagnostic system - the Molecular Microscope® Diagnostic System (MMDx) that interprets biopsies in terms of their molecular phenotype, and combines the molecular and histopathological features of transplant biopsies, plus clinical and laboratory parameters, to create the first Integrated Diagnostic System. The MMDx developed first in kidney transplant biopsies because phenotypes are well established, will now be adapted to heart transplant endomyocardial biopsies (EMBs). The present study will develop a Reference Set of EMB, adapt the MMDx system to assess and report EMBs; and validate and refine this system in 900 unselected prospectively collected for clinical indications and a standard of care EMBs from North American and European Centers. In addition to demonstrating the real-time feasibility and potential value of this System in patient care, the study will develop and optimize a transparent and user-friendly reporting format to communicate this information to clinicians and obtain detailed feedback to improve its utility. We refine now our MMDx system using a new type of analysis (see primary outcome) and the resulting MMDx report. Currently, INTERHEART recruited 1912 biopsies from 1279 patients.

ELIGIBILITY:
Inclusion Criteria:

* biopsy for clinical indications

Exclusion Criteria:

* no consent
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study aims to recruit 1200 biopsies from heart transplant patients for clinical indications and the standard of care biopsies.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2016-01; Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Assign molecular scores (probability) of T cell mediated rejection, antibody mediated rejection in heart transplant biopsies, in a reference set of 200 biopsies | 2 years
  Create a molecular classifier that predicts antibody mediated and T cell mediated rejection, based on the archetypal analysis.

SECONDARY OUTCOMES:
Assign in real time (three working days upon biopsy receipt) molecular scores (probability) of T cell mediated rejection and antibody mediated rejection. | 1 year
  The molecular phenotype of a newly acquired sample predicts the histologic and clinical features of this sample when compared to the reference set.

CONTACTS AND LOCATIONS:
Overall Officials: Philip F Halloran, MD PhD, Principal Investigator — University of Alberta
Locations (13):
- United States (5):
  - UCLA Medical Centre, Los Angeles, California
  - Cedars-Sinai Heart Institute, Los Angeles, California
  - Annette C. and Harold C. Simmons Transplant Institute, BaylorScott&White Research Institute, Dallas, Texas
  - Cardiovascular Medicine, University of Utah Health, Salt Lake City, Utah
  - Virginia Commonwealth University, Division of Cardiology, Richmond, Virginia
- Cardiac Transplantation Laboratory, The Victor Chang Cardiac Research Institute, Darlinghurst, Australia
- Department of Cardiac Surgery, Medical University of Vienna, Vienna, Austria
- Canada (2):
  - Alberta Transplant Applied Genomics Center, University of Alberta, Edmonton, Alberta
  - Division of Cardiology, University of Alberta, Edmonton, Alberta
- Institute for Clinical and Experimental Medicine - IKEM, Prague, Czechia
- Service de Néphrologie-Dialyse Adultes , Hôpital Necker-Enfants Malades, Paris, France
- Heart Failure and Heart Transplant Unit, University of Bologna, Bologna, Italy
- Advanced Heart Failure Transplant Unit, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Madill-Thomsen KS, Halloran PF. Precision diagnostics in transplanted organs using microarray-assessed gene expression: concepts and technical methods of the Molecular Microscope(R) Diagnostic System (MMDx). Clin Sci (Lond). 2024 Jun 5;138(11):663-685. doi: 10.1042/CS20220530. PMID 38819301
- [Result] Loupy A, Duong Van Huyen JP, Hidalgo L, Reeve J, Racape M, Aubert O, Venner JM, Falmuski K, Bories MC, Beuscart T, Guillemain R, Francois A, Pattier S, Toquet C, Gay A, Rouvier P, Varnous S, Leprince P, Empana JP, Lefaucheur C, Bruneval P, Jouven X, Halloran PF. Gene Expression Profiling for the Identification and Classification of Antibody-Mediated Heart Rejection. Circulation. 2017 Mar 7;135(10):917-935. doi: 10.1161/CIRCULATIONAHA.116.022907. Epub 2017 Feb 1. PMID 28148598
- [Result] Halloran PF, Potena L, Van Huyen JD, Bruneval P, Leone O, Kim DH, Jouven X, Reeve J, Loupy A. Building a tissue-based molecular diagnostic system in heart transplant rejection: The heart Molecular Microscope Diagnostic (MMDx) System. J Heart Lung Transplant. 2017 Nov;36(11):1192-1200. doi: 10.1016/j.healun.2017.05.029. Epub 2017 May 29. PMID 28662985
- [Result] Halloran PF, Reeve J, Aliabadi AZ, Cadeiras M, Crespo-Leiro MG, Deng M, Depasquale EC, Goekler J, Jouven X, Kim DH, Kobashigawa J, Loupy A, Macdonald P, Potena L, Zuckermann A, Parkes MD. Exploring the cardiac response to injury in heart transplant biopsies. JCI Insight. 2018 Oct 18;3(20):e123674. doi: 10.1172/jci.insight.123674. PMID 30333303
- [Result] Parkes MD, Aliabadi AZ, Cadeiras M, Crespo-Leiro MG, Deng M, Depasquale EC, Goekler J, Kim DH, Kobashigawa J, Loupy A, Macdonald P, Potena L, Zuckermann A, Halloran PF. An integrated molecular diagnostic report for heart transplant biopsies using an ensemble of diagnostic algorithms. J Heart Lung Transplant. 2019 Jun;38(6):636-646. doi: 10.1016/j.healun.2019.01.1318. Epub 2019 Feb 6. PMID 30795962
- [Result] Halloran PF, Madill-Thomsen KS. The Molecular Microscope Diagnostic System: Assessment of Rejection and Injury in Heart Transplant Biopsies. Transplantation. 2023 Jan 1;107(1):27-44. doi: 10.1097/TP.0000000000004323. Epub 2022 Dec 8. PMID 36508644
- [Result] Halloran PF, Madill-Thomsen K, Mackova M, Aliabadi-Zuckermann AZ, Cadeiras M, Crespo-Leiro MG, Depasquale EC, Deng M, Gokler J, Hall SA, Kim DH, Kobashigawa J, Macdonald P, Potena L, Shah K, Stehlik J, Zuckermann A, Reeve J. Molecular states associated with dysfunction and graft loss in heart transplants. J Heart Lung Transplant. 2024 Mar;43(3):508-518. doi: 10.1016/j.healun.2023.11.013. Epub 2023 Nov 30. PMID 38042442
- [Result] Halloran PF, Madill-Thomsen K, Aliabadi-Zuckermann AZ, Cadeiras M, Crespo-Leiro MG, Depasquale EC, Deng M, Gokler J, Kim DH, Kobashigawa J, Macdonald P, Potena L, Shah K, Stehlik J, Zuckermann A. Many heart transplant biopsies currently diagnosed as no rejection have mild molecular antibody-mediated rejection-related changes. J Heart Lung Transplant. 2022 Mar;41(3):334-344. doi: 10.1016/j.healun.2021.08.004. Epub 2021 Aug 26. PMID 34548198
- [Result] Halloran PF, Madill-Thomsen K, Aliabadi-Zuckermann AZ, Cadeiras M, Crespo-Leiro MG, Depasquale EC, Deng M, Gokler J, Hall S, Jamil A, Kim DH, Kobashigawa J, Macdonald P, Melenovsky V, Patel J, Potena L, Shah K, Stehlik J, Zuckermann A. Redefining the molecular rejection states in 3230 heart transplant biopsies: Relationships to parenchymal injury and graft survival. Am J Transplant. 2024 Aug;24(8):1414-1426. doi: 10.1016/j.ajt.2024.03.031. Epub 2024 Mar 26. PMID 38527588
- [Derived] Madill-Thomsen KS, Reeve J, Aliabadi-Zuckermann A, Cadeiras M, Crespo-Leiro MG, Depasquale EC, Deng M, Goekler J, Kim DH, Kobashigawa J, Macdonald P, Potena L, Shah K, Stehlik J, Zuckermann A, Halloran PF. Assessing the Relationship Between Molecular Rejection and Parenchymal Injury in Heart Transplant Biopsies. Transplantation. 2022 Nov 1;106(11):2205-2216. doi: 10.1097/TP.0000000000004231. Epub 2022 Oct 21. PMID 35968995
- [Derived] Halloran PF. Integrating molecular and histologic interpretation of transplant biopsies. Clin Transplant. 2021 Apr;35(4):e14244. doi: 10.1111/ctr.14244. Epub 2021 Feb 17. No abstract available. PMID 33595110